CLINICAL TRIAL: NCT04546672
Title: An Assessor-blinded, Randomized, Controlled, Single Center, Parallel Design Trial With Patient Masking to Compare Early Postoperative Gastric Emptying Associated With Rocuronium Neuromuscular Reversal With Sugammadex Versus Neostigmine in Adults Undergoing Colon and Rectal Surgery
Brief Title: Sugammadex To IMprove Bowel Function
Acronym: STIM_Bowel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Brandon M Togioka, Director of Clinical Research-Anesthesiology, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 21895; MISP #60224 (Other Grant/Funding Number: Merck & Co., INC.)
Record Dates: First submitted 2020-09-05; First posted 2020-09-14 (Actual); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Bowel Dysfunction; Postoperative Complications; Neuromuscular Blockade
Keywords: sugammadex; neostigmine; Gastric emptying; neuromuscular blockade
MeSH Terms: conditions — Intestinal Diseases; Postoperative Complications | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Intervention Model Description: Assessor-blinded, randomized, controlled, single center, parallel design trial with patient masking
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sugammadex (Experimental): Sugammadex 2 mg/kg IV once at the end of surgery
  Interventions: Drug: Sugammadex
- Neostigmine (Active Comparator): Neostigmine 0.07 mg/kg to a maximum of 5 mg (+Glycopyrrolate 0.2 mg per 1 mg of neostigmine administered) IV once at the end of surgery
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex — At the end of the surgical procedure at a depth of neuromuscular blockade after the reappearance of T2 on the train-of-four, Sugammadex will be dosed once at 2 mg/kg actual body weight through an intravenous line with brisk flow
  Other Names: Org 25969; Bridion
  Arms: Sugammadex
Drug: Neostigmine — At the end of surgical procedure at a depth of neuromuscular blockade after the reappearance of T2 on the train-of-four, Neostigmine will be dosed once at 0.07 mg/kg actual body weight to a maximum of 5 mg through an intravenous line with brisk flow. Glycopyrrolate will be coadministered with Neostigmine at a dose of 0.2 mg of Glycopyrrolate per 1.0 mg of Neostigmine administered
  Other Names: Prostigmin; Vagostigmin
  Arms: Neostigmine

SUMMARY:
Colon and rectal surgery is associated with high cost, long length of stay, high postoperative surgical site infection rate, high incidence of postoperative nausea and vomiting, and a high rate of hospital readmission. Return of bowel function is of utmost importance in avoiding patient discomfort, morbidity, and mortality after colorectal surgery. All patient having colorectal surgery receive neuromuscular paralysis, which is reversed at the end of surgery with either glycopyrrolate and neostigmine, or sugammadex. Glycopyrrolate and neostigmine both affect bowel function. Sugammadex has no effect on bowel function. The purpose of this study is to determine if a strategy of neuromuscular reversal with sugammadex, instead of glycopyrrolate and neostigmine, may increase gastric emptying after surgery and lead to less postoperative complications.

DETAILED DESCRIPTION:
Colon and rectal surgery is associated with high cost, long length of stay, high postoperative surgical site infection rate, high incidence of postoperative nausea and vomiting, and a high rate of hospital readmission. The 30-day mortality rate after open or laparoscopic surgery for colorectal cancer is high-between 3 and 8%. Return of bowel function is of utmost importance in avoiding patient discomfort, morbidity, and mortality after colorectal surgery. The incidence of postoperative ileus after colorectal surgery has been reported to be 10-25%. Postoperative ileus is defined as intolerance of oral intake due to a lack of coordinated bowel motility. Significant attention has been paid to the development of guidelines and programs to reduce the incidence of postoperative ileus and accelerate return of bowel function after colorectal surgery.

The American Society of Colon and Rectal Surgeons (ASCRS) and the Society of American Gastrointestinal and Endoscopic Surgeons (SAGES) created an enhanced recovery after surgery (ERAS) protocol to promote the following outcomes in patients undergoing colorectal surgery: "freedom from nausea, freedom from pain at rest, early return of bowel function, improved wound healing, and early hospital discharge". An intervention that facilitates faster postoperative gastric emptying may impact many of these outcomes; in particular, nausea may be reduced, constipation-associated pain at rest may decline, return of bowel function would be accelerated, and time to hospital discharge may be shortened. While administration of medications such as Alvimopan and adjustments in anesthetic technique (providing epidural analgesia, minimizing crystalloid administration, using multimodal analgesia) are recommended, sugammadex is not currently considered in the ERAS protocol.

Neuromuscular paralysis is required for the duration of open and laparoscopic colorectal surgery to decrease patient movement, improve operating conditions, and at times facilitate ventilation. Neostigmine and glycopyrrolate are commonly used to reverse rocuronium neuromuscular blockade at the end of surgery. Both neostigmine and glycopyrrolate impact bowel function. Neostigmine promotes and glycopyrrolate slows gastrointestinal motility. Co-administration of neostigmine and glycopyrrolate can have variable effects on return of bowel function after surgery. In general, administering a higher proportion of neostigmine than glycopyrrolate is associated with faster return of bowel function. Unopposed cholinergic activity from neostigmine administration can cause morbidity including bradycardia, bronchoconstriction, hypotension, urinary incontinence, and increased salivary secretions. Thus, the ratio of neostigmine to glycopyrrolate is relatively fixed and cannot be adjusted to promote desired gastrointestinal outcomes. Sugammadex does not bind to acetylcholine receptors on bowel and is presumed not to affect bowel function.

Some investigations into the contribution of sugammadex versus acetylcholinesterase inhibitors to recovery of bowel function have been completed. In retrospective studies, sugammadex administration has been associated with faster time to first bowel movement and less ileus-related delays in hospital discharge. Conversely, two randomized, controlled clinical trials found no difference in outcomes related to gastrointestinal motility including time to first flatus, time to first bowel movement, and incidence of postoperative ileus. One randomized, controlled trial found a shorter time to first flatus, but no difference in time to first bowel movement. Lastly, one study found a trend towards faster gastric emptying with sugammadex. A limitation of the aforementioned prospective studies is they include patients having surgery on their thyroid gland, gallbladder, and other intraabdominal organs. These surgeries lack bowel handling and anastomosis, which translates to less effect on postoperative bowel function. It is hypothesized that a randomized, controlled trial involving patients having colorectal surgery will find faster gastric emptying, less nausea, and less gastrointestinal complications (including ileus) when sugammadex is administered to reverse rocuronium neuromuscular blockade, compared to neostigmine.

The purpose of this study is to determine if administering sugammadex for reversal of neuromuscular blockade instead of neostigmine and glycopyrrolate, a strategy that avoids cholinergic effects on the bowel, is associated with faster gastric emptying, faster time to achieve a TOFr > 0.9, less post-surgical gastrointestinal complications, shorter time to first bowel movement, shorter PACU phase 1 recovery, and shorter hospital length of stay. If sugammadex is shown to improve the aforementioned outcomes, an argument can be made that sugammadex should be considered for inclusion in the ERAS protocol for Colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Having surgery in the South Operating Rooms at Oregon Health & Science University
* Surgery scheduled Monday through Friday
* Having colorectal surgery
* Planned general endotracheal anesthesia

Exclusion Criteria:

* Prisoners
* Pregnant women
* An inability to consent for surgery or anesthesia
* Allergy to a study drug
* Medical contraindication to neuromuscular blockade
* Stage 4 kidney disease or worse (glomerular filtration rate < 30 ml/min)
* Significant liver dysfunction (Aspartate transaminase or Alanine transaminase > twice the OHSU normal)
* Taking Toremifene

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon M Togioka, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Togioka BM, Rakshe SK, Ye S, Tekkali P, Tsikitis VL, Fang SH, Herzig DO, Lu KC, Aziz MF. A Randomized Controlled Trial of Sugammadex versus Neostigmine for Reversal of Rocuronium on Gastric Emptying in Adults Undergoing Elective Colorectal Surgery. Anesth Analg. 2025 Aug 1;141(2):373-383. doi: 10.1213/ANE.0000000000007518. Epub 2025 May 6. PMID 40327558

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sugammadex | Neostigmine
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex | Neostigmine | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (13.2) | 55.9 (14.0) | 56.4 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 55
  Male | 31 | 34 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 59 | 58 | 117
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 57 | 55 | 112
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.2 (9.6) | 28.1 (6.4) | 28.6 (8.2)
ASA Physical Status [Count of Participants; unit: Participants]
  1-normal health | 0 | 2 | 2
  2-mild systemic disease | 22 | 25 | 47
  3-severe systemic disease | 38 | 32 | 70
  4-severe systemic disease that is a constant threat to life | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Gastric Emptying
Description: Gastric emptying as assessed by the area under the paracetamol concentration-time curve by trapezoidal approximation (AUC)
Time Frame: 150 minutes after neuromuscular reversal
Measure: Mean (Standard Deviation); unit: log(ng*ml-1)*min
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 60 | 60
log(ng*ml-1)*min | 1120 (122) | 1130 (117)
Statistical Analysis 1: Comparison: Sugammadex vs Neostigmine; Test type: Superiority; p = 0.58, t-test, 2 sided; Mean Difference (Final Values) = 12.1, 95% CI 2-sided [-31.1 to 55.4]

2. Secondary Outcome: Time in Minutes to Reach Train of Four (TOF) Ratio ≥ 0.9 After the Administration of Reversal Drug.
Description: The TOF ratio will be measured in continuous manner every 15 seconds after the administration of reversal drug. The TOF ratio will be measured by the TwitchView electromyograph. The TOF ratio was measured in this study by stimulating the ulnar nerve with four equal stimuli at a frequency of 2 hertz. The TOF ratio is calculated by dividing the amplitude of the muscle response from the fourth stimuli by the amplitude of the muscle response from the first stimuli.
Time Frame: 30 minutes after the administration of reversal drug.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 60 | 60
minutes | 5.2 (6.3) | 17.5 (10.1)
Statistical Analysis 1: Comparison: Sugammadex vs Neostigmine; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 12.3, 95% CI 2-sided [9.2 to 15.4]

3. Secondary Outcome: Number of Participants With Gastrointestinal Complications
Description: Gastrointestinal complications will include all of the following: anastomotic leak, postoperative ileus, reoperation, and organ space infection. National Surgical Quality Improvement Project definitions will be used. Active monitoring for these outcomes will occur on an ongoing daily basis until hospital discharge. In addition, chart review and patient phone call will occur 30 days after discharge to assess for complications after discharge.
Time Frame: 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 60 | 60
Participants | 10 | 19
Statistical Analysis 1: Comparison: Sugammadex vs Neostigmine; Test type: Superiority; p = 0.087, Fisher Exact; Odds Ratio (OR) = 2.3, 95% CI 2-sided [0.9 to 6.2]

4. Secondary Outcome: PACU Recovery Time
Description: The time to attain pain control and stable respiratory, hemodynamic, and neurologic status after surgery.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 60 | 60
minutes | 115 (50.3) | 108 (56.4)
Statistical Analysis 1: Comparison: Sugammadex vs Neostigmine; Test type: Superiority; p = 0.48, t-test, 2 sided; Mean Difference (Final Values) = -6.9, 95% CI 2-sided [-26.4 to 12.6]

5. Secondary Outcome: Reversal Time to First Bowel Movement
Description: The time from reversal of neuromuscular blockade to first bowel movement
Time Frame: length hospitalization, an average of 1 week
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 60 | 60
hours | 44.3 (33.8) | 61 (43)
Statistical Analysis 1: Comparison: Sugammadex vs Neostigmine; Test type: Superiority; p = 0.02, t-test, 2 sided; Mean Difference (Final Values) = 16.7, 95% CI 2-sided [2.3 to 31.1]

6. Secondary Outcome: Reversal Time to Discharge Order
Description: The number of days between reversal of neuromuscular blockade and time of discharge order
Time Frame: length of hospitalization, an average of 1 week
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 60 | 60
days | 4.8 (4.9) | 7.82 (19.8)
Statistical Analysis 1: Comparison: Sugammadex vs Neostigmine; Test type: Superiority; p = 0.27, t-test, 2 sided; Mean Difference (Final Values) = 3, 95% CI 2-sided [-2.2 to 8.3]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Sugammadex | Neostigmine
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 2/60 | 5/60
Other Adverse Events (participants affected / at risk) | 10/60 | 13/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex (N=60) | Neostigmine (N=60)
Hypersensitivity Reaction (Immune system disorders) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Upper Airway Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex (N=60) | Neostigmine (N=60)
nausea or vomiting (Gastrointestinal disorders) | 7 (7) | 10 (10)
Foul, salty, or metallic taste (Nervous system disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/72/NCT04546672/Prot_SAP_000.pdf